CLINICAL TRIAL: NCT07240506
Title: Effect of Acute Caffeine Intake Via Caffeinated Gum on Vertical Jump Performance in Female Volleyball Players: A Single-Blind Placebo-Controlled Trial
Brief Title: Effect of Caffeinated Chewing Gum on Vertical Jump Performance in Female Volleyball Players
Acronym: CAF-GUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muttalip Ayar (Other)
Responsible Party: Sponsor-Investigator, Muttalip Ayar, Assistant Professor, University of Beykent
Organization: University of Beykent (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: E-10840098-202.3.02-735
Record Dates: First submitted 2025-11-16; First posted 2025-11-21 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Athletic Performance
Keywords: Caffeine; Caffeinated Gum; Female Athletes; Jump Performance; Sports Nutrition

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeinated Gum (CAF) (Experimental): Participants chewed two pieces of caffeinated chewing gum containing a total of 200 mg caffeine (2 × 100 mg). After chewing for 5 minutes, they performed squat jump, countermovement jump, and block jump tests.
  Interventions: Dietary Supplement: Caffeinated chewing gum
- Placebo Gum (PLA) (Placebo Comparator): Participants chewed two pieces of placebo chewing gum identical in appearance and flavor but containing no caffeine. After chewing for 5 minutes, they performed the same vertical jump tests as in the caffeinated condition.
  Interventions: Dietary Supplement: Placebo chewing gum

INTERVENTIONS:
Dietary Supplement: Caffeinated chewing gum — Two pieces of caffeinated chewing gum providing 200 mg total caffeine; administered 15 minutes before performance testing.
  Arms: Caffeinated Gum (CAF)
Dietary Supplement: Placebo chewing gum — Two pieces of placebo chewing gum identical in appearance and flavor to the caffeinated gum but containing no caffeine; administered 15 minutes before performance testing.
  Arms: Placebo Gum (PLA)

SUMMARY:
This study aimed to examine the acute effects of caffeine intake through caffeinated chewing gum on the vertical jump performance of professional female volleyball players. Ten athletes from the Turkish Women's Volleyball First League voluntarily participated in this single-blind, placebo-controlled, randomized crossover study. Each athlete completed two test sessions: one with caffeinated gum containing 200 mg of caffeine and one with a caffeine-free placebo gum. After chewing the gum for 5 minutes, participants performed three types of vertical jump tests: squat jump, countermovement jump, and block jump. The results showed that caffeinated gum significantly improved countermovement jump height compared with the placebo, while no significant differences were observed for squat or block jumps. The findings suggest that caffeine in gum form may enhance explosive performance in sports requiring rapid power output, such as volleyball.

DETAILED DESCRIPTION:
Caffeine is a well-established ergogenic aid known to improve endurance, strength, and cognitive performance. However, limited evidence exists on its acute effects in female team-sport athletes. This study was designed to evaluate the impact of acute caffeine intake via caffeinated chewing gum on vertical jump performance among professional female volleyball players. The research employed a randomized, single-blind, placebo-controlled crossover design.

Ten professional athletes aged 18-33 years from the Yeşilyurt Sports Club Women's A Team, competing in the Turkish Volleyball Federation Women's 1st League, were included. Participants underwent two experimental sessions: one involving caffeinated gum (CAF, 200 mg total caffeine from two 100 mg pieces) and one involving placebo gum (PLA, identical but caffeine-free), separated by a six-day washout period. The gums were chewed for 5 minutes, and jump performance tests were conducted 15 minutes later.

Vertical jump performance was evaluated using a Chronojump jump mat for three jump types: squat jump (SJ), countermovement jump (CMJ), and block jump (BJ). Each test included three attempts, with the highest score recorded for analysis. Data were analyzed with paired-sample t-tests using SPSS 27.0, with significance set at p<0.05.

The results showed that caffeine gum significantly increased CMJ height compared with the placebo (p<0.05), but no significant effects were observed for SJ or BJ performance. The findings indicate that caffeine in gum form may acutely improve explosive performance involving stretch-shortening cycle movements.

The study was approved by the Non-Interventional Clinical Research Ethics Committee of Istanbul Medipol University (Approval No: E-10840098-202.3.02-735). All participants provided informed consent prior to data collection.

ELIGIBILITY:
Inclusion Criteria:

Self-identified female athletes aged 18-33 years Professional volleyball players actively competing in the Turkish Women's Volleyball First League Minimum of 3 years of competitive volleyball experience Healthy individuals without any diagnosed medical conditions Willing to abstain from caffeine-containing products for at least 24 hours before each testing session Voluntarily agreed to participate and provided written informed consent

Exclusion Criteria:

Known cardiovascular, metabolic, or neurological disorders Current use of medications or supplements affecting physical performance or caffeine metabolism Pregnancy or breastfeeding History of caffeine sensitivity, intolerance, or allergy Failure to comply with pre-test instructions (e.g., caffeine restriction, rest period) Musculoskeletal injuries preventing full jump performance

Ages: 18 Years to 33 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only self-identified female athletes were eligible to participate in this study. Participants were professional volleyball players competing in the Turkish Women's Volleyball First League.
Enrollment: 10 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Countermovement Jump Height | Within 15 minutes after gum administration.
  Change in countermovement jump (CMJ) height measured using a Chronojump contact mat following caffeine or placebo gum ingestion.

SECONDARY OUTCOMES:
Squat Jump Height | Within 15 minutes after gum administration.
  Change in squat jump (SJ) height measured using a Chronojump contact mat after caffeine or placebo gum ingestion.
Block Jump Height | Within 15 minutes after gum administration.
  Change in block jump (BJ) height measured using a Chronojump contact mat after caffeine or placebo gum ingestion.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeşilyurt Sports Club - Women's Volleyball Team Training Facility, Istanbul, Bakırköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset contains identifiable information related to a small group of professional athletes. Only summarized results are available within the published manuscript and supplementary materials upon reasonable request.